CLINICAL TRIAL: NCT03509857
Title: Vibration Analgesia in Propofol Infusion During Anesthesia Induction
Acronym: VAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Aravind Pothula, Principal investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-8323
Record Dates: First submitted 2018-01-04; First posted 2018-04-26 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pain, Acute
Keywords: Pain; Acute pain; Analgesia; Propofol infusion
MeSH Terms: conditions — Acute Pain; Pain; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- normal standard of care infusion of propofol without analgesia (Placebo Comparator): normal standard of care infusion of propofol without analgesia
  Interventions: Other: No Intervention
- infusion of propofol with application of vibration analgesia (Experimental): infusion of propofol with application of vibration analgesia
  Interventions: Device: BUZZY(tm)

INTERVENTIONS:
Device: BUZZY(tm) — Risks associated with the BUZZY(tm) device The intervention group will receive vibration only, with application of the BUZZY device just proximal to the intravenous infusion site immediately before and during propofol infusion.
  There are no known risks for the use of the BUZZY(tm) device, which is registered as an FDA class III device ("therapeutic massager").
  Arms: infusion of propofol with application of vibration analgesia
Other: No Intervention — No intervention
  Arms: normal standard of care infusion of propofol without analgesia

SUMMARY:
In this study, the investigators seek to evaluate the role of vibration in the reduction of discomfort associated with painful stimulus associated with anesthesia induction. Through this study, the investigators hope to develop a comprehensive and cost-effective approach to minimize patient discomfort during anesthesia induction.

DETAILED DESCRIPTION:
Background and Significance Infusion of propofol during the process of inducing anesthesia can cause a fair amount of transient discomfort to patients while the are on the operating table and of intact faculties. It is not uncommon for patients to cry out in pain. The investigators have noticed this first hand on numerous occasions and have wondered if there is a risk-free way to lesson the pain associated with propofol infusion.

This study will focus on the use of vibration analgesia to potentially reduce the pain associated with propofol infusion. Vibration is proposed to stimulate A-beta nerve fibers, which transmit information from vibration and touch which, according to the Gate Control Theory of Pain (Melzack and Wall 1965), inhibits signal transduction by A-delta and C fibers (Kakigi and Shibasaki 1992). Vibration has been demonstrated to be effective to decrease pain during vaccinations, phlebotomy, and dental anesthesia (Baxter et al. 2011; Nanitsos et al. 2009).

In this study, the investigators seek to evaluate the role of vibration in the reduction of discomfort associated with painful stimulus associated with anesthesia induction. Through this study, the investigators hope to develop a comprehensive and cost-effective approach to minimize patient discomfort during anesthesia induction.

Study Design

The objective of this study is to evaluate the effectiveness of vibration as a analgesic during induction of anesthesia. It is the investigators hypothesis that both vibration will lessen the pain of propofol infusion.

Patients set to receive a propofol infusion as part of induction of anesthesia during surgery will be recruited to participate in this study. All participating patients will be randomized following acquisition of consent for study participation to one of two intervention groups: 1) normal standard of care infusion of propofol without analgesia 2) infusion of propofol with application of vibration analgesia. Patients will then be asked to place a mark on a 100-mm visual analogue scale corresponding to the level of pain that they experienced during the digital block. Additionally, Please see the next section for specific details regarding the intervention.

Due to constraints regarding the validity of the linear visual analogue scale in very young patients (Stinson et al. 2006), only those aged 18 years or older will be eligible for participation in the study. Parents or guardians will provide consent for minors or for individuals who are otherwise unable to provide consent themselves.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 to 100 who are going to receive propofol injection as part of induction of anesthesia for surgery

Exclusion Criteria:

* Those below the age of 18

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aravind Pothula, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Hutchinson Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baxter AL, Cohen LL, McElvery HL, Lawson ML, von Baeyer CL. An integration of vibration and cold relieves venipuncture pain in a pediatric emergency department. Pediatr Emerg Care. 2011 Dec;27(12):1151-6. doi: 10.1097/PEC.0b013e318237ace4. PMID 22134226
- [Background] Bini G, Cruccu G, Hagbarth KE, Schady W, Torebjork E. Analgesic effect of vibration and cooling on pain induced by intraneural electrical stimulation. Pain. 1984 Mar;18(3):239-248. doi: 10.1016/0304-3959(84)90819-4. PMID 6203084
- [Background] Depue K, Christopher NC, Raed M, Forbes ML, Besunder J, Reed MD. Efficacy of intravenous lidocaine to reduce pain and distress associated with propofol infusion in pediatric patients during procedural sedation. Pediatr Emerg Care. 2013 Jan;29(1):13-6. doi: 10.1097/PEC.0b013e31827b227e. PMID 23283255
- [Background] Grauers A, Liljeroth E, Akeson J. Propofol infusion rate does not affect local pain on injection. Acta Anaesthesiol Scand. 2002 Apr;46(4):361-3. doi: 10.1034/j.1399-6576.2002.460405.x. PMID 11952433
- [Background] Kakigi R, Shibasaki H. Mechanisms of pain relief by vibration and movement. J Neurol Neurosurg Psychiatry. 1992 Apr;55(4):282-6. doi: 10.1136/jnnp.55.4.282. PMID 1583512
- [Background] Lee JR, Jung CW, Lee YH. Reduction of pain during induction with target-controlled propofol and remifentanil. Br J Anaesth. 2007 Dec;99(6):876-80. doi: 10.1093/bja/aem293. PMID 18006530
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Nanitsos E, Vartuli R, Forte A, Dennison PJ, Peck CC. The effect of vibration on pain during local anaesthesia injections. Aust Dent J. 2009 Jun;54(2):94-100. doi: 10.1111/j.1834-7819.2009.01100.x. PMID 19473149
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: normal standard of care infusion of propofol without analgesia
- Treatment Group: Infusion of propofol with vibration analgesia
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Greater than 18
  years | 51.5 (14.2) | 50 (13.7) | 50.7 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 20 | 20 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — New York, USA
  participants
    United States | 50 | 50 | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — BMI
  kg/m^2 | 30.9 (9.3) | 29.4 (5.2) | 30.2 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain as Observed by Two Independent Observers Following Propofol Injection, With or Without a Vibration Analgesia Adjunct
Description: Patient pain will be assessed by two independent observers, an attending anesthesiologist and a certified registered nurse anesthetist (CRNA). Pain was graded using a four-point pain manifestation scale described by McCrirrick & Hunter : 0 = none (negative response to questioning), 1 = mild (pain reported in response to questioning only, without any behavioral signs), 2 = moderate (pain reported in response to questioning and accompanied by a behavioral sign, or pain reported spontaneously without questioning), 3 = severe (strong vocal response or response accompanied by facial grimacing, arm withdrawal or tears). Higher scores meaning worse outcome (perceived pain) and lower score meaning better outcome.
Time Frame: Day 1 at time of propofol injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 50 | 50
units on a scale | 3.1 (1.6) | 1.4 (0.5)

ADVERSE EVENTS:
Time Frame: Up to 1 month following post-operative treatment.
Description: The risks related to vibration therapy is minimal
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03509857/Prot_003.pdf
  • Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03509857/SAP_004.pdf
  • Informed Consent Form (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03509857/ICF_005.pdf